CLINICAL TRIAL: NCT07087444
Title: The Effectiveness of Health Education Intervention in Enhancing Personal Protective Equipment and Visibility Material Use Among Commercial Motorcycle Riders and Passengers in the Limbe and Tiko Health District of Cameroon
Brief Title: The Effectiveness of Health Education Intervention in Enhancing Personal Protective Equipment Use
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Buea (Other)
Collaborators: University of California, Los Angeles (Other); University of California, Berkeley (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Chrisantus Eweh Ukah, PhD Fellow / Principal Investigator, University of Buea
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2490-03; D43TW012186 (NIH)
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Road Traffic Injury Prevention, Motorcycle Safety, Personal Protective Equipment Use, Visibility Materials, Injury Prevention Education, Health Behavior Change
Keywords: Motorcycle safety, personal protective equipment, visibility materials, road injury prevention, health education, commercial riders, Cameroon, road safety
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment design involving two groups: the intervention group in Limbe Health District, which receives a health education program to improve uptake of personal protective equipment (PPE) and visibility materials, and the control group in Tiko Health District, which does not receive the intervention during the study period. Both groups are followed simultaneously to compare changes in knowledge, attitudes, and use of safety equipment. Participants are commercial motorcycle riders and passengers aged 18 years and above. This design allows assessment of the effectiveness of the health education intervention by comparing outcomes between intervention and control communities.
Masking Description: No masking (open-label) was implemented in this study. Participants, care providers, investigators, and outcomes assessors were aware of group assignments due to the nature of the health education intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 Title: Intervention Group (Limbe Health District) (Experimental): Participants in the Limbe Health District receive a structured health education intervention designed to improve their knowledge, attitudes, and use of personal protective equipment (PPE) and visibility materials. The intervention includes interactive group sessions, distribution of educational materials, and follow-up reminders via SMS to reinforce safe riding practices. This aims to increase the consistent use of helmets, reflective jackets, and other visibility aids to reduce road traffic injuries among commercial motorcycle riders and passengers.
  Interventions: Behavioral: Health education intervention to improve knowledge and uptake of personal protective equipment and visibility materials among commercial motorcycle riders and passengers
- Arm 2 Title: Control Group (Tiko Health District) (No Intervention): Participants in the Tiko Health District serve as the control group and do not receive the health education intervention during the study period. They continue their usual practices without additional education or support related to personal protective equipment or visibility materials. This allows comparison to assess the effectiveness of the intervention delivered in Limbe.

INTERVENTIONS:
Behavioral: Health education intervention to improve knowledge and uptake of personal protective equipment and visibility materials among commercial motorcycle riders and passengers — This intervention consists of a structured health education program targeting commercial motorcycle riders and passengers in the Limbe Health District. It includes interactive group sessions focused on the importance, benefits, and correct use of personal protective equipment (helmets, reflective jackets) and visibility materials (reflective strips, lights). Educational materials such as leaflets and posters are distributed to reinforce learning. Additionally, participants receive follow-up SMS reminders to encourage consistent and proper use of protective gear. The goal is to increase awareness and uptake of safety measures to reduce road traffic injuries. This intervention is community-based and tailored to the local context in Cameroon.
  Arms: Arm 1 Title: Intervention Group (Limbe Health District)

SUMMARY:
This study is testing whether a health education program can help commercial motorcycle riders and passengers in the Limbe and Tiko Health Districts of Cameroon improve their use of safety equipment. These include items like helmets, reflective jackets, and other materials that help riders and passengers be more visible and protected on the road.

People who ride or travel on motorcycles are at high risk for road injuries, especially when visibility is low. Wearing personal protective equipment (PPE) and visibility materials can prevent many of these injuries, but many riders do not use them regularly.

The study involves educating riders and passengers through group sessions and follow-up messages about the importance of safety gear. We will compare the use of PPE and visibility materials before and after the health education intervention to see if it made a difference.

Adults aged 18 and older who ride or travel on motorcycles in Limbe or Tiko are eligible to participate. The study will last several months and does not involve any drugs or medical procedures. There is no known risk to participants.

The results will help guide future road safety programs in Cameroon and other similar settings

DETAILED DESCRIPTION:
Commercial motorcycle riders and passengers in Cameroon face a high burden of road traffic injuries, especially in crisis-affected areas like the Limbe and Tiko Health Districts. Poor road visibility, limited use of personal protective equipment (PPE), and low awareness of road safety practices contribute significantly to these injuries.

Despite the known benefits of PPE such as helmets, reflective jackets, and visibility materials, their uptake remains low. Previous studies have shown that health education can improve safety behaviors, but there is limited evidence on its effectiveness in increasing the use of PPE and visibility materials in this high-risk population.

This study aims to assess the impact of a targeted health education intervention on the uptake of PPE and visibility materials among commercial motorcycle riders and passengers. The intervention includes interactive education sessions, distribution of educational materials, and follow-up communication through SMS. Participants' knowledge, attitudes, and use of safety equipment will be measured before and after the intervention to evaluate effectiveness.

The findings from this study will support the design of scalable and community-driven road safety interventions and may inform national policy and programming to reduce road traffic injuries in Cameroon and similar low-resource settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and above

Commercial motorcycle riders or regular motorcycle passengers

Residing or operating in the Limbe or Tiko Health District

Willing and able to provide informed consent

Able to participate in both baseline and follow-up assessments

Exclusion Criteria:

* Individuals who declined to provide informed consent

Individuals who were not available for follow-up or unwilling to participate in follow-up assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 967 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Uptake of personal protective equipment and visibility materials | From enrollment to endline at 6 months
  Change in the proportion of motorcycle riders and passengers reporting consistent use of PPE (helmets, reflective jackets) and visibility materials (reflective strips, lights) before and after the intervention.

SECONDARY OUTCOMES:
Change in knowledge level on the importance of PPE and visibility materials | 6 months
  Improvement in participants' knowledge scores (based on a structured questionnaire) about the role of PPE and visibility materials in road safety.
Change in attitudes toward use of PPE and visibility materials | Baseline and 6 months post-intervention
  Improvement in participants' attitude scores toward the regular and appropriate use of PPE and visibility materials.

CONTACTS AND LOCATIONS:
Overall Officials: Chrisantus Eweh Ukah, PhD Fellow, Principal Investigator — UNIVERSITY OF BUEA, Cameroon
Locations (1):
- University of Buea, Buea, SWR, Cameroon

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the study will be made available after de-identification. Data will be shared with researchers who provide a methodologically sound proposal and agree to use the data only for research purposes. Data will be available starting 6 months after publication and for up to 5 years. To request access, contact the Principal Investigator at [your email].
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication and 5 years after the start date
Access Criteria: Individual participant data (IPD) and supporting documents will be accessible to qualified researchers who submit a scientifically sound research proposal related to the study objectives. Researchers must agree to use the data solely for research purposes and to maintain participant confidentiality. Access will be granted after approval by the Principal Investigator or the study steering committee. Data and documents will be shared via secure data transfer methods upon signing a data use agreement. Requests can be submitted by contacting the Principal Investigator at chrisantuseweh@gmail.com.
URL: https://www.ubuea.cm

REFERENCES:
- [Background] Ukah CE, Tendongfor N, Hubbard A, Tanue EA, Oke R, Bassah N, McCoy SI, Yunika LK, Ngu CN, Hemono R, Christie SA, Nsagha DS, Chichom-Mefire A, Juillard C. Knowledge and attitudes of commercial motorcyclists on personal protective equipment in the crisis-affected Limbe and Tiko Health Districts of Cameroon toward injury prevention: A formative research study for a health education intervention. medRxiv [Preprint]. 2025 May 7:2025.05.06.25327113. doi: 10.1101/2025.05.06.25327113. PMID 40385440
- See also: Preprint of the study on knowledge and attitudes of commercial motorcyclists regarding personal protective equipment in Limbe and Tiko Health Districts, Cameroon, available on medRxiv. — https://www.medrxiv.org/content/10.1101/2025.05.06.25327113v1